CLINICAL TRIAL: NCT04072744
Title: Foot Oedema Observed Over Time in Heart Failure Patients
Brief Title: Foot Oedema Observed Over Time Study
Acronym: FOOT
Status: Completed | Type: Observational
Sponsor: Heartfelt Technologies (Industry)
Collaborators: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TSD01
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Edema Leg
Keywords: Peripheral oedema; Peripheral edema; Heart failure; Decompensation; Weight; Hospital admissions
MeSH Terms: conditions — Heart Failure; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: General Study Participants
  Interventions: Device: Heartfelt measurements; Device: Connected weighing scales

INTERVENTIONS:
Device: Heartfelt measurements — The measurements taken using the Heartfelt device do not require contact with the participant. For the measurements to take place, the participant will simply walk in the field of view of the device. As the device(s) will have been installed at a location allowing the best view of where the participant goes in an out of bed, the participant is not expected to change anything to their routine.
  The device can also take measurements in the dark, so if the participant walks in front of the device in the dark, this information will also be captured.
  The Heartfelt device is a CE (European Conformity) marked product. Neither the participant, or the medical team will be able to see the data collected by the Heartfelt device during the study. They will be blinded to the data until each participant has completed the study. At that point they can choose to review the data from participant individually or wait until all the data from all participants is available.
Device: Connected weighing scales — The participant will be instructed to use those scales for the period of the study, as often as directed by their healthcare professional. The weighing scales display weight so that the participants can record the weight in their own heart failure records.
  The participant will be able to see the weight readings on the weighing scales during the study.
  The scales will communicate with the Personal Computer (PC) contained in the Heartfelt device and the data will be sent to the Heartfelt server through an encrypted link.

SUMMARY:
Heart Failure is the final common pathway of most forms of cardiovascular disease. In the United Kingdom (UK), it affects around 900 000 people, causes or complicates around 5% of adult emergency hospital admissions and consumes up to 2% of total National Health Service (NHS) expenditure. An important part of discharge planning includes measures such as early follow up in order to prevent readmissions. The hallmark of heart failure is fluid retention and between 2009 and 2016, 43% to 50% of hospital admissions were associated with peripheral oedema. Therefore, early recognition of this and treatment of the congestion may prevent hospital admissions. In clinical trials, management strategies have included patient education, telemedicine and remote monitoring. The main non-invasive method for detecting fluid retention has been the use of weight as a surrogate marker.

The Heartfelt device is an invention that uses a system of cameras in a compact device in order to generate 3 dimensional images of the feet and lower legs. The volumes can then be calculated and thus, changes in amount of peripheral oedema can be estimated. In a laboratory study performed by the Heart Failure team at the Royal Brompton Hospital, there was good correlation between measurements made by Heartfelt and a water displacement method. The resolution was as good as 20mls.

By positioning the Heartfelt device in the bedroom, automatic measurements can be made whenever the subject gets in and out of bed. Images are only taken of the specified subject. Data is censored so that the part of the body which is 50cm above the floor is not stored. Encrypted, anonymised data is transmitted over the internet to the company's secure servers. Personal identifiable data (participant name, address, age…) is stored on an encrypted hard drive, along with linkage information (device serial numbers) to associate the participant identifiable data with the data captured in the home. Therefore, data collection is not only secure but entirely passive, which is a major advantage compared with previous non-invasive methods and it is applicable to a very wide range of compliant and non-compliant patients.

Our hypothesis is that the Heartfelt device can directly detect the increase in peripheral oedema associated with heart failure decompensation and that, on average, the number of days with missing data collected by the Heartfelt device will be lower than that of the weighing scales.

DETAILED DESCRIPTION:
This is a phase 2 observational study during which Subjects with chronic heart failure will be monitored in their home using the Heartfelt device.

The participant inclusion criteria will be those patients who are at high risk of hospital admission with a primary diagnosis of chronic heart failure or pulmonary oedema due to Heart failure (HF), during either of which peripheral oedema was also noted.

When heart failure decompensates, the amount of peripheral oedema that is clinically significant is unknown. The main objective of this study is to characterise the volume changes indicative of an increased risk for subsequent hospitalisation.

Subjects will also be provided with electronic, internet connected weighing scales that can transmit data and asked to weigh themselves daily. Temporal changes in weight and volume will be compared.

The study period will be 6 months and is the interval between installation of the Heartfelt device and the study end. participants will be made aware that the data collected by the device will not be reviewed during the study and therefore that they should continue with reporting symptoms and issues as usual to their care team.

In the event that it takes more than 2 years to recruit 20 participants, the study team will stop recruiting after 2 years so the study will be considered complete when all participants recruited up to that point have been monitored for 6 months.

participants under the care of the Trust have the following post diagnosis care:

* Patient Education and Training in self management

  * Daily weighing
  * Diuretic management
* Discharged under cardiologist
* Home visit by heart failure nurse (HFN) at 7-10d
* Urgent contact info for HF team
* Subsequent HF care by

  * HFN either at home or at community hospital
  * Consultant cardiologist

The Heartfelt Device will be provided in addition to these and not replace any of these activities.

During the study period, data will be collected from the Heartfelt device (passively) and a set of connected weighing scales (as and when the participant steps on the scales). Any decisions made by the subject to seek medical help will not be influenced by the research team or the Heartfelt device readings as those would be concealed to the participant and research team until appropriate review during the study. The participant will however be able to see the readings on the weighing scales as they step on it.

Retrospective analysis of the participant's notes which may indicate change in medications or care will be mapped to the foot volumes and weights collected.

For those participants for whom decompensation occurs during the study period, the participants are seen by their healthcare professionals, and a clinical examination will be made as usual in a timely manner to determine the amount of peripheral oedema. This will be logged allowing retrospective comparison with the volume measurements.

The temporal relationship between volume changes and decompensation will be investigated. The additional effect of clinical status data will be assessed.

As the participation in a scientific study is known to modify behaviour, the information collected by scales and general reporting frequency of symptoms will be compared to the 6 months before the study and the 6 months after. The time to recruit participants should correct for any seasonal effect on this data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years or older.
2. Patient able, agrees and signs the Informed Consent Form.
3. Patient with any heart failure diagnosis.
4. Patient under the care of a cardiologist with heart failure nurse care.
5. Patient with one prolonged inpatient stay
6. Patient with significant peripheral oedema at admission
7. Patient with significant weight loss following admission (at least 5kg weight loss).
8. Patient has been discharged on at least furosemide 80mg or Bumetanide 2mg/d

Exclusion Criteria:

1. Patient has bandages everyday
2. Patient has an amputation of the foot
3. Patient lacks capacity to consent
4. Patient is of no fixed abode
5. Patient has plans for intervention (CRT, Valves)
6. Patient taking part in another study
7. Patient must not been pregnant, and is taking relevant birth control*

   * Note that criteria (g) has been requested by the insurance for clinical trial cover. However we do not expect participants of this study to be trying to get pregnant (participants are expected to be over 55 years old).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Locally resident patients who are under the care of the cardiology / heart failure team with a high risk for heart failure related hospital admission, are potentially eligible.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in foot volume prior to Heart failure related hospital admission | Through study completion, an average of 6 months
  The primary outcome is the change in foot volume between baseline and the last observed foot volume measurement prior to hospital admission for a given patient. This will aim to demonstrate the ability of the heartfelt system to provide advance warning of impending hospitalisation.

SECONDARY OUTCOMES:
Frequency of data collection by the Heartfelt Device | Through study completion, an average of 6 months
  the frequency with which the heartfelt system collects patient data in comparison to standard care (weighing scales).
Correlation between foot volume and significant medical intervention | Through study completion, an average of 6 months
  The correlation between the dates of significant medical interventions (change of diuretics, hospital admission...) and difference in foot volumes to baseline measured by the Heartfelt device.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Keeling, MD, Principal Investigator — Torbay and South Devon NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Bedfordshire Hospitals NHS Foundation Trust, Luton, Bedfordshire
  - North Tees and Hartlepool Hospitals NHS Foundation Trust, Stockton-on-Tees, County Durham
  - Torbay and South Devon NHS Foundation Trust, Torquay, Devon
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Northumbria Healthcare NHS Foundation Trust, North Shields, Northumbria

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with other researchers